# A MOBILE PHONE SHORT MESSAGE SERVICE INTERVENTION TO INCREASE RETENTION IN HIV CARE AMONG HIV-POSITIVE MEN WHO HAVE SEX WITH MEN (MSM) IN PERU

#### **WELTEL PERU**

#### **SUMMARY**

Retention in care (or in care) for HIV is associated with increased survival and viral suppression, and with less transmission of the virus. HIV disproportionately affects men who have sex with men (MSM). In Peru, the HIV epidemic is concentrated in them (prevalence of 12.2%), while only 0.4% of the general population is HIV+. What is concerning is that MSM tend to have lower rates of retention in HIV care. Studies with text messages (SMS) have been reported to be effective in promoting testing for HIV and other sexually transmitted infections in MSM. Two-way text messaging (2-way, ie when the patient can reply) can provide a higher level of real-time support to patients. WelTel was the first randomized controlled trial to use this interactive approach and reported a significant increase in adherence and viral suppression. WelTel has been used successfully for HIV, asthma and tuberculosis. However, further studies are needed to evaluate the use of this strategy to increase retention in HIV care in resource-limited settings, such as in Latin America. The hypothesis is that an adapted version of WelTel can be used to implement a 2-way text message-based intervention, and to increase retention in care among HIV+ MSM in Peru.

To address the low retention in HIV care among MSM in Lima, we will use the WelTel system and its strategy managed by health providers consisting of sending reminder and informative SMS and differentiated follow-up. We will assess the efficacy of the intervention with a randomized controlled trial comparing the proportion of HIV+ MSM retained in HIV care among those who received the intervention versus the standard care arm, up to one year after enrollment. We will recruit 208 participants who will be randomly assigned (1:1) to an intervention group (receives the intervention with WelTel) and a control group (standard of care). Delivery of the intervention will take place over 6 months, and the main outcome to be measured will be retention in HIV care up to 1 year after enrollment.

#### **ACRONYM**

PLWHA: people living with HIV/AIDS. MSM: men who have sex with men.

ART: antiretroviral therapy.

SMS: short message service (short text message).

CD4: CD4 T lymphocyte cell.

CV: viral load. RR: relative risk.

MINSA: Ministry of Health.

PS: health provider.

STIs: sexually transmitted infections.

#### RESEARCHERS

Dr. Luis Menacho Dr. Giovani Díaz Dra. Magaly Blas Dra. Elsa Gonzáles

#### INTRODUCTION

23.3 million people living with HIV/AIDS (PLWHA) are now receiving antiretroviral therapy (ART) and it is estimated that there will be 2.8 million more per year in the next 3 years (19). For continued access to ART and monitoring of clinical and virological progress, PLWHA must be maintained in high-quality care. **Retention in HIV care is associated with increased survival, viral suppression; and reduced HIV transmission and viral resistance** (20,21). Missing more than two HIV care visits increased mortality risk in a multicenter cohort study (HR = 3.61; 95% CI, 2.35-5.55) (21). Low retention in HIV care is a critical barrier to achieving optimal individual and community outcomes. Continuum of HIV care includes testing for exclusion, linkage to care, initiation of ART, retention, and adherence to therapy to achieve and maintain viral suppression. Since 2010, the number of new HIV infections in Latin America has remained stable, without significant decreases as observed in all other regions of the world (19). Viral suppression remains low in some regions: 22% in the Middle East and North Africa; 40% in the Caribbean; and 52% in Latin America (19). With the expansion of ART, urgent efforts are needed to retain PLWHA in care and thus reduce morbidity, mortality, and the incidence of new HIV-related infections (22-24).

HIV disproportionately affects men who have sex with men (MSM). MSM represent 41% of new infections in the region (19). In fact, MSM have a 27-fold higher risk of HIV infection than the general population (25). In Peru, the epidemic is concentrated among them (prevalence 12.2%), while only 0.4% of the general population is HIV+ (19,26). The incidence among MSM aged 18 to 29 years has increased substantially and 60% of new infections occur in this group (27,28). Of concern, HIV-positive MSM are less likely to remain in care than other population groups (29-33). In the United States, 54.3% retention in HIV care and 50.8% viral suppression were reported among MSM aged 20-24 years (32). In Peru, less than 50% of MSM have been tested for HIV and it is estimated that only 24% of those infected know their status (28). The Ministry of Health reported that retention in HIV care after the first year is 55%, which drops significantly during the second year (26). National viral suppression is only 36% (26).

Based on multiple studies that have shown efficacy, the World Health Organization (WHO) strongly recommends the use of text messages (mobile health) to improve adherence to ART (34-38). However, evidence on the impact of mobile health for retention in HIV care is scarce (39,40). Some studies in Africa concluded that short message service reminders (SMS or text messages) are effective in improving retention in HIV care in the general population (39). Until now, no controlled study has done the same with MSM, one of the populations most affected by HIV. Studies with MSM have reported good efficacy of SMS reminders to promote testing for HIV

and other sexually transmitted infections (STIs) (41-43). More trials with this key population are needed to evaluate the use of SMS to increase retention in HIV care in resource-limited settings, such as in Latin America (39).

Two-way communication (between patient and healthcare provider) with text messages (SMS) has the potential to provide comprehensive care through improved communication. A meta-analysis comparing one-way versus two-way SMS found that two-way SMS is the main driver for improving treatment adherence, while one-way messages have little or no benefit (44). Two-way messaging can provide a higher level of real-time support to patients. An evaluation of this strategy using the "behavior change wheel" suggested that the flow of support after an initial SMS is a key contributor to improving ART adherence (45). Health providers need appropriate tools to optimize the delivery of two-way text-based interventions and make them feasible and easy to deliver (38). An existing tool supported by evidence from previous studies can be adapted for use with MSM in Peru, with the aim of optimizing the delivery of a two-way text message intervention to increase retention in HIV care (38).

**WelTel** was the first randomized controlled trial using an interactive two-way text messaging approach that reported a significant increase in adherence and viral suppression in Kenya (RR for non-adherence: 0.81, 95% CI: 0.69 -0.94; RR for virologic failure 0.84, 95% CI: 0.71-0.99), as well as among HIV+ women in Vancouver, BC (38,46). WelTel is based on a well-structured platform that connects healthcare providers with patients through regular text messages. It uses a web-based program (software) (accessed through the Internet) with intuitive functionalities that allow providers to monitor, track and support large numbers of people (47). The platform allows addressing multiple morbidities, as well as different health services. The system has been tested in Kenya, Rwanda, South Africa, the United States, and Canada and has been used for other diseases such as tuberculosis and asthma (46,48,49). A recent study with WelTel in Kenya significantly improved Quality of Life scores ("the 4th 90") (40). HIV+ MSM in Peru may benefit from receiving an SMS-based intervention delivered through the WelTel platform to increase low retention in HIV care (retention = 50% at study site).

#### **JUSTIFICATION**

Peru is a relevant place to test an SMS intervention to increase retention in HIV care based on existing WelTel technology. The country has a high number of cell phone subscriptions (121 per 100 people), and smartphone use is also very common and constantly growing (50-52). Our preliminary data shows that Peruvian MSM are interested in receiving HIV prevention information via SMS (2,3,50,53). Other studies report that HIV+ MSM are interested in interacting with health providers to discuss HIV-related issues that may positively affect their retention in care (55). The proposed study will develop, implement, and evaluate an adapted version of WelTel to deliver a two-way interactive SMS intervention to increase retention among HIV+ MSM. WelTel has been used extensively in other resource-limited settings, and there is preliminary information in Peru to help tailor the content of such an intervention (3,4,12,40,43,49,55).

The use of a two-way SMS intervention to improve retention in HIV care among MSM is innovative. Globally, there are no published controlled studies on improving retention among HIV+ MSM that have used this approach and this study will be the first to evaluate this type of mHealth intervention in Peru. This study will provide evidence on the use of mobile health to improve retention in HIV care, where retention is currently very low. Retention has been the focus of fewer interventions compared to other steps of the HIV care continuum, and it is a crucial step because it involves multiple visits over time (35,57-59). This is the first study that will test the WelTel system in Latin America, specifically in Peru, where there are promising characteristics to carry out the intervention. We will adapt and validate the system for use in Spanish. We will test an already developed system that has the flexibility to add new features to improve patient follow-up.

#### **OBJECTIVES**

# **General Objective:**

To assess the efficacy of a text message (SMS)-based strategy delivered with the support of a web tool (WelTel) to increase retention in HIV care in Peru.

# **Specific Objective:**

To determine the efficacy of SMS-based intervention delivered through the WelTel system in increasing retention in HIV care compared to standard care.

# **Hypothesis:**

An SMS-based intervention delivered through the WelTel system will increase retention in HIV care among MSM. We hope to increase retention in HIV care from 50% to 70%.

### **METHODS**

#### **Study Overview:**

To address the low retention in HIV care among MSM in Lima, we will use the WelTel system and its strategy managed by health providers that consists of sending reminder and informative SMS and with differentiated follow-up. We will assess the efficacy of the intervention with a randomized controlled trial comparing the proportion of HIV+ MSM retained in HIV care versus the standard care arm up to one year after enrollment. Table 1 summarizes the exposures, results, and design.

#### **Behavior Theory:**

The <u>behavior change wheel framework</u> has been used to explain how WelTel can promote adherence to ART. The Capability, Opportunity, Motivation, and Behavior model is at the core of the theory (45). According to this model, the achievement of a behavior requires the presence of capacity, opportunity and motivation. To perform in a behavior, a person needs psychological (knowledge and skills) and physical capacity. Opportunity (physical and social) refers to factors that promote behavior. Physical opportunities are those that occur in the external environment, such as a physical reminder (SMS) to take medication. Social opportunities refer to non-physical factors, such as social norms and interpersonal influences. Motivation includes automatic and

reflexive processes that elicit behaviors such as emotions, habits, beliefs, and plans. Automatic processes are those that involve emotional responses, impulses, desires, and reflex responses, while reflective processes involve conscious planning and evaluation. This framework advocates identifying behavior change techniques as components of the intervention.

Only 1 behavior change technique has been identified for the automated text messaging component of the intervention: requesting/indicating the behavior. The behavior change techniques identified in WelTel were mainly related to its personalized communication component delivered to patients who reported a problem or query. These techniques were: a) eliciting/indicating the behavior, b) unspecified social support, c) reducing negative emotions, d) communication from a credible source, e) information about health consequences, f) social emotional support, g) practical social support, eh) instructions on how to perform a behavior. At WelTel, such behavior change techniques were linked to 5 intervention functions: environmental restructuring, empowerment, education, persuasion, and training.

Finally, to specify possible mechanisms of action to promote a behavior, such techniques and functions must be connected to influences on behavior following this model. The proposed mechanisms of action to facilitate adherence behavior in WelTel were: a) the delivery of an external trigger (SMS reminder to complete a behavior) and social support, to influence opportunities and automatic motivation through restructuring and environmental clearance; b) delivery of health-related information and social support to influence ability, opportunity, and motivation through education, persuasion, and training. We believe that retention in HIV care will be similarly influenced in our intervention.

# **General description:**

This intervention will be designed for MSM who are HIV positive. We will recruit subjects 18 years of age or older. The intervention will begin one day after enrollment. The two-way SMS intervention will have four components: 1) an automated weekly SMS sent to ask how they are doing (basic follow-up); 2) phone calls from a health provider to participants who respond that they have a problem, or that they need support or some information that cannot be resolved by text message; 3) SMS reminder 1 week before an appointment for HIV care.

#### Design:

Randomized controlled trial.

# **Main result:**

The primary outcome will be retention in HIV care for up to 1 year after enrollment. Participants will be classified as retained in care if they attend three HIV care appointments that are separated by 90 days or more within a one-year period (at the study HIV center) (64). Otherwise, they will be classified as not retained. The delivery of the intervention will last 6 months and the follow-up period to verify retention will last up to 12 months.

# Main exposure:

Text message (SMS) based intervention delivered through the WelTel system by trained health providers.

#### **Procedures:**

- 1. **Recruitment and eligibility criteria**. We will identify and recruit 208 HIV+ MSM in the Cayetano Heredia Hospital HIV service for a period of up to 12 months. <u>Eligible participants</u> will be 1) men who have sex with men; 2) 18 years or older; 3) has been diagnosed HIV positive; 4) own a cell phone that can send and receive SMS; 5) resides in Lima; and 6) not be enrolled in another study that uses text messaging.
- 2. Enrollment and randomization: During enrollment, the recruiter will be blinded to assignment to the intervention group. The recruiter will obtain informed consent and instruct the participant on how he should interact if he starts receiving text messages (see appendix 1). Participants will be randomly assigned after providing their cell phone number and brief general information (first name, date of diagnosis, email). They will be assigned a study ID and randomly divided into intervention or control arm (1:1 ratio) using computer generated random numbers. Arm assignments will be in sequentially numbered sealed envelopes. Healthcare providers trained to administer the intervention will be informed by the research team when a new participant is enrolled in the intervention arm. Due to the nature of the study, healthcare providers and participants will not be blinded to group assignment. The participants assigned to the intervention arm will have their telephone numbers registered on the platform.
- 3. Intervention. We will use the WelTel platform. For 6 months, every Monday the system will send automatic SMS with the question "How are you?" or similar questions (How are you?; How are you doing?). Participants will be instructed to respond if they are okay ("All OK") or if they have a problem ("I want support"; "I'm not okay"). The provider will send a return SMS to participants who have a problem or query; or they will call those who need it. The WelTel program has a customizable dictionary that identifies the words (or phrases) that the administrator indicates; thus, the answers of the participants are automatically ordered to indicate who needs follow-up through a reply SMS or call. One week before each appointment for HIV care, health providers will send an SMS reminder (Table 1).
- 4. Standard care arm. In 2018, the government published new national guidelines for HIV care (65). After pre-test counseling, the diagnosis of HIV is made with two rapid tests. Those who test positive for both tests receive post-test counselling, including emotional support, and are linked to an ART initiation center, ideally within the same week. During the first medical appointment after diagnosis, laboratory tests including CD4 and viral load (VL) are requested. In most cases, initiation of antiretroviral treatment (ART) occurs at the second medical appointment when basic laboratory results are available. Currently, it is not mandatory to have CD4/CV results available to start ART. ART, viral load and CD4

lab tests are provided free of charge. It is recommended that patients have CD4 counts and viral load testing twice during the first year. A one-month supply of ART is initially provided. If patients are adherent, nurses dispense ART every 3 months and also assess adherence.

Table 1. Summary of the study: exposures, results and design.

| Component | Sub- | Description |
|---|---|---|
| | component | |
| | Basic follow-up | Weekly automatic SMS with the question "How are you?" or similar |
| | SMS (check-in) | messages. This will be shipped for 6 months. |
| Intervention | Calls | The provider can call participants who have a problem. |
| arm | Appointment | SMS reminder one week before each appointment for HIV care. |
| (exposure) | reminders | |
| | Primary | Retention in HIV care up to 1 year after enrollment, defined as attending 3 |
| Results | | appointments that are 90 days apart within a 1-year period. |
| | Desing | Randomized controlled trial with a parallel group. |
| | | We aim to increase retention in HIV care from 50% to 70%. With 104 |
| | Sample size | participants in each arm, we will have 80% power to detect this difference |
| Design | Follow-up | 6 months (intervention); 12 months (retention measure). |
| | Theory | The behavior change wheel framework and its model of Capability, |
| | | Opportunity, Motivation and Behavior. |
| | Standard of care | Post-test counselling, including emotional support and linkage to ART |
| Control arm | | initiation, ideally within a week. ART, CD4, and viral load laboratory tests are |
| | | provided free of charge in Peru. |

#### Analysis plan:

 Data sources for the main result. The main outcome to be measured will be retention in HIV care during the first year after enrollment. Retention in care will be considered if they attend 3 HIV care appointments that are at least 90 days apart within a one-year period (64). We will verify retention in HIV care with: study registration (enrollment) sheets, physical medical records from the HIV service, reception appointment notebooks, and with a final follow-up survey.

Health providers will enter the data from the enrollment registration sheets into a database that will be stored in a password-protected computer file. The data from the final follow-up online survey completed by the participants will be exported to the physical database and will be periodically deleted from the online survey system server. All data resulting from the interaction between providers and participants will be stored on the WelTel platform that has high security standards: encrypted, password protected and HIPAA compliant (*The Health Insurance Portability and Accountability Act*).

Statistic analysis. for the main outcome, we will compare the proportion of MSM who
were retained in care in both groups, as a cumulative incidence rate. If any variable of
interest is not balanced between intervention and control arms, we will calculate Mantel

Haenszel-adjusted relative risks (RR). For secondary outcomes, we will also assess differences in the proportion of participants.

3. **Calculation of the sample size**. We hope to increase retention in HIV care from 50% to 70% one year after enrollment in the study clinic among HIV+ MSM. With 104 participants in each arm, we will have 80% power to detect this difference.

Our main outcome is the degree of loss to follow-up. Retention in care at the study HIV service (as opposed to being lost to follow-up) is the primary outcome, and retention in any HIV clinic will be a secondary measure. Participants lost to follow-up will be considered as not retained. We will measure the retention in an establishment of the Ministry of Health (MINSA). MINSA provides care to more than 60% of Peruvians (73). Since retaining subjects in our public health system is an important goal, we have not adjusted the sample size calculation based on the potential loss of subjects to follow-up.

#### **OPERATIONALIZATION OF VARIABLES**

**Table 2**. Operationalization of variables.

| Variable | Туре | Options | Source |
|---|---|---|---|
| Age | Continuous | > 18 | Online follow-up survey |
| Education | Categorical | Secondary, Technical,<br>Superior, | Online follow-up survey |
| Civil status | Categorical | Single, Married,<br>Outgoing, Coupled | Online follow-up survey |
| Employment situation | | | Online follow-up survey |
| Nationality | | | Online follow-up survey |
| sexual orientation | exual orientation Categorical | | Online follow-up survey |
| Diagnosis date | Date | Day month Year | Clinic history; dating record |
| Treatment start date | Date | Day month Year | Clinic history; dating record |
| Attended appointment dates | Date | Day month Year | Clinic history; dating record |
| Viral load | Continuous | | Clinic history |
| CD4 | Continuous | | Clinic history |
| alcohol use | numeric | | Online follow-up survey |
| Condom use, last encounter | Categorical | Yes, No | Online follow-up survey |
| Email | Text | | enrollment sheet |
| Cell phone number | Numeric | NA | enrollment sheet |
| Arm | Categorical | Control, Intervention | Study Database |
| Retention in HIV care | Categorical | If not; Attend three appointments for HIV care that are 90 days or more apart within a one-year period (at the study HIV center) | Clinic history; dating<br>record; online follow-up<br>survey; WelTel system |

#### TIMELINE

| Actividades | | Year 1 | | | Year 2 | | | Year 3 | | | Year 4 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 |
| Recruitment/Enrollment | | | | | | | | | | | | | | | | |
| Delivery of intervention | | | | | | | | | | | | | | | | |
| Monitoring and analysis | | | | | | | | | | | | | | | | |
| Manuscript development | | | | | | | | | | | | | | | | |

#### REFERENCES

- 1. Huisa BN, Menacho LA, Rodriguez S, Bustos JA, Gilman RH, Tsang VC, Gonzalez AE, García HH; Cysticercosis Working Group in Peru. Taeniasis and cysticercosis in housemaids working in affluent neighborhoods in Lima, Peru. Am J Trop Med Hyg. 2005 Sep;73(3):496-500.
- 2. Menacho L, Garcia PJ, Blas MM, Díaz G, Zunt JR. What Men Who Have Sex With Men in Peru Want in Internet-Based Sexual Health Information. J Homosex. 2018;65(7):934-946. doi: 10.1080/00918369.2017.1364939. Epub 2017 Sep 22.
- 3. Blas MM, Menacho LA, Alva IE, Cabello R, Orellana ER. Motivating men who have sex with men to get tested for HIV through the internet and mobile phones: a qualitative study. PLoS One. 2013;8(1):e54012.
- 4. Menacho LA, Blas MM, Alva IE, Roberto Orellana E. Short Text Messages to Motivate HIV Testing Among Men Who have Sex with Men: A Qualitative Study in Lima, Peru. Open AIDS J. 2013 Apr 5;7:1-6.
- Chiu CJ, Menacho L, Young SD. The Association Between Age and Ethics-Related Issues in Using Social Media for HIV Prevention in Peru. Ethics Behav. 2016;26(2):99-109.
- 6. Young SD, Cumberland WG, Nianogo R, Menacho LA, Galea JT, et al. The HOPE social media intervention for global HIV prevention in Peru: a cluster randomised controlled trial. The lancet HIV. 2015 January; 2(1):27-32.
- 7. Menacho LA, Galea JT, Young SD. Feasibility of Recruiting Peer Educators to Promote HIV Testing Using Facebook Among Men Who have Sex with Men in Peru. AIDS Behav. 2015 Jun;19 Suppl 2:123-9.
- 8. Krueger EA, Chiu CJ, Menacho LA, Young SD. HIV testing among social media-using Peruvian men who have sex with men: correlates and social context. AIDS Care. 2016 Oct;28(10):1301-5.

- 9. Garett R, Menacho L, Young SD. Ethical Issues in Using Social Media to Deliver an HIV Prevention Intervention: Results from the HOPE Peru Study. Prev Sci. 2017 Feb;18(2):225-232.
- 10. Young SD, Nianogo RA, Chiu CJ, Menacho L, Galea J. Substance use and sexual risk behaviors among Peruvian MSM social media users. AIDS Care. 2016;28(1):112-8.
- 11. Blas MM, Brown B, Menacho L, Alva IE, Silva-Santisteban A, Carcamo C. HPV Prevalence in Multiple Anatomical Sites among Men Who Have Sex with Men in Peru. PLoS One. 2015 Oct 5;10(10):e0139524.
- 12. Bayona E, Menacho L, Segura ER, Mburu G, Roman F, Tristan C, Bromley E, Cabello R. The Experiences of Newly Diagnosed Men Who Have Sex with Men Entering the HIV Care Cascade in Lima, Peru, 2015-2016: A Qualitative Analysis of Counselor-Participant Text Message Exchanges. Cyberpsychol Behav Soc Netw. 2017 Jun;20(6):389-396.
- 13. WhatsApp as a tool to support recently diagnosed gay men with HIV in Peru. International Association of Providers of AIDS Care (IAPAC) conference June 2017. Oral presentation. Retrieved from: https://www.iapac.org/AdherenceConference/presentations/ADH2017 OA244.pdf
- 14. Barriers and facilitators of HIV care in recently diagnosed men who have sex with men (MSM) in Lima, Peru: qualitative analysis of bi-directional text messages from an mHealth intervention. International AIDS society (IAS) conference July 2017. Poster. Retrieved from: http://programme.ias2017.org/Abstract/Abstract/5233
- 15. Video "Victor": developed for improving linkage to HIV care among recently diagnosed men who have sex with men at Via Libre that can be seen at https://www.youtube.com/watch?v=7H1CGzIYro4&t=20s; presented at International AIDS society conference 2016: http://programme.aids2016.org/Programme/Session/899
- 16. Video "Differentiated service delivery for adolescents": developed as an e-learning strategy to improve the HIV continuum of care. Retrieved from: https://www.youtube.com/watch?feature=share&v=eFiDSkncoUE&app=desktop
- 17. Lama JR, Brezak A, Dobbins JG, Sanchez H, Cabello R, Rios J, Bain C, Ulrich A, De la Grecca R, Sanchez J, Duerr A. Design Strategy of the Sabes Study: Diagnosis and Treatment of Early HIV Infection Among Men Who Have Sex With Men and Transgender Women in Lima, Peru, 2013-2017. Am J Epidemiol. 2018 Mar 7.
- 18. Menacho LA, Blas MM. [How to produce a video to promote HIV testing in men who have sex with men?]. Rev Peru Med Exp Salud Publica. 2015 Jul-Sep;32(3):519-25.
- 19. UNAIDS data 2018. Retrieved from: http://www.unaids.org/sites/default/files/media asset/unaids-data-2018 en.pdf
- 20. Giordano TP, Gifford AL, White AC Jr, et al. Retention in care: a challenge to survival with HIV infection. Clin Infect Dis 2007; 44:1493–9.
- 21. Mugavero MJ, Westfall AO, Cole SR, Geng EH, Crane HM, et al. Centers for AIDS Research Network of Integrated Clinical Systems (CNICS). Beyond core indicators of

- retention in HIV care: missed clinic visits are independently associated with all-cause mortality. Clin Infect Dis. 2014 Nov 15;59(10):1471-9.
- 22. Govindasamy D, Kranzer K, Ford N. Strengthening the HIV cascade to ensure an effective future ART response in sub-Saharan Africa. Trans R Soc Trop Med Hyg. 2014 Jan;108(1):1-3.
- 23. Granich RM, Gilks CF, Dye C et al. Universal voluntary HIV testing with immediate antiretroviral therapy as a strategy for elimination of HIV transmission: a mathematical model. Lancet 2009;373:48–57.
- 24. Rebeiro PF, Cesar C, Shepherd BE, De Boni RB, Cortés CP, et al. Assessing the HIV Care Continuum in Latin America: progress in clinical retention, cART use and viral suppression. J Int AIDS Soc. 2016 Apr 8;19(1):20636.
- 25. UNAIDS 2018 Global HIV Statistics. Fact Sheet Global AIDS Update 2019. Retrieved from: http://www.unaids.org/sites/default/files/media asset/UNAIDS FactSheet en.pdf
- 26. Garcia-Fernandez L, Novoa R, Huaman B, Benites C. Continuum of care of people living with HIV and gaps in achieving the 90-90-90 goals in Peru. Rev Peru Med Exp Salud Publica. 2018;35(3):491-6.
- 27. Epidemiological situation of HIV-AIDS in Peru. National Center for Epidemiology, Prevention and Control of Diseaseskk, Peruvian Ministry of Health. Monthly Bulletin, June 2018. Retrieved from: <a href="http://www.dge.gob.pe/portal/docs/vigilancia/vih/Boletin\_2018/junio.pdf">http://www.dge.gob.pe/portal/docs/vigilancia/vih/Boletin\_2018/junio.pdf</a>
- 28. Chow JY, Konda KA, Borquez A, Caballero P, Silva-Santisteban A, et al. Peru's HIV care continuum among men who have sex with men and transgender women: opportunities to optimize treatment and prevention. Int J STD AIDS. 2016 Oct;27(12):1039-1048.
- 29. Castro R, Ribeiro-Alves M, Corrêa RG, Derrico M, Lemos K, et al. The Men Who Have Sex with Men HIV Care Cascade in Rio de Janeiro, Brazil. PLoS One. 2016 Jun 14;11(6):e0157309.
- 30. Hussen SA, Harper GW, Bauermeister JA, Hightow-Weidman LB. Psychosocial influences on engagement in care among HIV-positive young black gay/bisexual and other men who have sex with men. AIDS Patient Care STDS. 2015 Feb; 29(2):77–85.
- 31. Hightow-Weidman L, Muessig K, Knudtson K, Srivatsa M, Lawrence E, LeGrand S, et al. A Gamified Smartphone App to Support Engagement in Care and Medication Adherence for HIV-Positive Young Men Who Have Sex With Men (AllyQuest): Development and Pilot Study. JMIR Public Health Surveill. 2018 Apr 30;4(2):e34.
- 32. Singh S, Mitsch 1, Wu B. HIV Care Outcomes Among Men Who Have Sex With Men With Diagnosed HIV Infection United States, 2015. MMWR Morb Mortal Wkly Rep. 2017 Sep 22;66(37):969-974.
- 33. Tanner AE, Mann L, Song E, Alonzo J, Schafer K, et al. weCARE: A Social Media-Based Intervention Designed to Increase HIV Care Linkage, Retention, and Health

- Outcomes for Racially and Ethnically Diverse Young MSM. AIDS Educ Prev. 2016 Jun;28(3):216-30.
- 34. Consolidated Guidelines on the Use of Antiretroviral Drugs for Treating and Preventing HIV Infection, 2nd edition. Recommendations for a Public Health Approach Geneva: World Health Organization; 2016. ISBN-13: 978-92-4-154968-4. Retrieved from: <a href="https://www.ncbi.nlm.nih.gov/books/NBK374294/">https://www.ncbi.nlm.nih.gov/books/NBK374294/</a>
- 35. Muessig KE, LeGrand S, Horvath KJ, Bauermeister JA, Hightow-Weidman LB. Recent mobile health interventions to support medication adherence among HIV-positive MSM.Curr Opin HIV AIDS. 2017 Sep;12(5):432-441.
- 36. Mayer JE, Fontelo P. Meta-analysis on the effect of text message reminders for HIV-related compliance. AIDS Care 2017; 29:409–417.
- 37. Kanters S, Park JJ, Chan K, et al. Interventions to improve adherence to antiretroviral therapy: a systematic review and network meta-analysis. Lancet HIV 2017; 4:e31–e40.
- 38. Lester RT, Ritvo P, Mills EJ, Kariri A, Karanja S, et al. Effects of a mobile phone short message service on antiretroviral treatment adherence in Kenya (WelTel Kenya1): a randomised trial. Lancet. 2010 Nov 27;376(9755):1838-45.
- 39. Jong S, Cuca Y, Thompson LM. Meta-analysis of Mobile Phone Reminders on HIV Patients' Retention to Care. J Mob Technol Med. 2017;6(1):5-18.
- 40. Van der Kop ML, Muhula S, Nagide PI, Thabane L, Gelmon L, Lester RT6 et al. Effect of an interactive text-messaging service on patient retention during the first year of HIV care in Kenya (WelTel Retain): an open-label, randomised parallel-group study. Lancet Public Health. 2018 Mar;3(3):e143-e152.
- 41. Bourne C, Knight V, Guy R, Wand H, Lu H, McNulty A. Short message service reminder intervention doubles sexually transmitted infection/HIV re-testing rates among men who have sex with men. Sex Transm Infect 2011 4;87(3):229–31.
- 42. Zou H, Fairley CK, Guy R, Bilardi J, Bradshaw CS, Garland SM, et al. Automated, Computer Generated Reminders and Increased Detection of Gonorrhoea, Chlamydia and Syphilis in Men Who Have Sex with Men.
- 43. Purnomo J, Coote K, Mao L, Fan L, Gold J, Ahmad R, Zhang L. Using eHealth to engage and retain priority populations in the HIV treatment and care cascade in the Asia-Pacific region: a systematic review of literature. BMC Infect Dis. 2018 Feb 17;18(1):82.
- 44. Wald DS, Butt S, Bestwick JP. One-way versus two-way text messaging on improving medication adherence: meta-analysis of randomized trials. Am J Med. 2015 Oct;128(10):1139.e1-5.
- 45. N, Guo M, Amico KR, Atkins L, Lester RT. Interactive Two-Way mHealth Interventions for Improving Medication Adherence: An Evaluation Using The Behaviour Change Wheel Framework. JMIR Mhealth Uhealth. 2018 Apr 12;6(4):e87.

- 46. King E, Kinvig K, Steif J, Qiu AQ, Maan EJ, et al. Mobile Text Messaging to Improve Medication Adherence and Viral Load in a Vulnerable Canadian Population Living With Human Immunodeficiency Virus: A Repeated Measures Study. J Med Internet Res. 2017 Jun 1;19(6):e190.
- 47. Lester RT1, Mills EJ, Kariri A, Ritvo P, Chung M, eta al. The HAART cell phone adherence trial (WelTel Kenya1): a randomized controlled trial protocol. Trials. 2009 Sep 22:10:87.
- 48. De Vera MA, Sadatsafavi M, Tsao NW, Lynd LD, Lester R, et al. Empowering pharmacists in asthma management through interactive SMS (EmPhAsIS): study protocol for a randomized controlled trial. Trials. 2014 Dec 13;15:488.
- 49. Van der Kop ML, Memetovic J, Patel A, Marra F, Sadatsafavi M, et al. The effect of weekly text-message communication on treatment completion among patients with latent tuberculosis infection: study protocol for a randomised controlled trial (WelTel LTBI). BMJ Open. 2014 Apr 9;4(4):e004362.
- 50. World Bank. Mobile cellular subscriptions. Retrieved from: <a href="https://data.worldbank.org/indicator/IT.CEL.SETS.P2">https://data.worldbank.org/indicator/IT.CEL.SETS.P2</a>
- 51. Gestion. Penetration of smartphones in Peru almost tripled in last four years. Retrieved from: <a href="https://gestion.pe/economia/empresas/penetracion-smartphones-peru-triplico-ultimos-cuatro-anos-225607">https://gestion.pe/economia/empresas/penetracion-smartphones-peru-triplico-ultimos-cuatro-anos-225607</a>
- 52. National Institute of Statistics and Informatics. Retrieved from: https://www.inei.gob.pe
- 53. Blas MM, Alva IE, Cabello R, Garcia PJ, Carcamo C, Redmon M, Kimball AM, Ryan R, Kurth AE. Internet as a tool to access high-risk men who have sex with men from a resource-constrained setting: a study from Peru. Sex Transm Infect. 2007 Dec;83(7):567-70.
- 54. Krishnan A, Ferro EG, Weikum D, Vagenas P, Lama JR, Sanchez J, Altice FL. Communication technology use and mHealth acceptance among HIV-infected men who have sex with men in Peru: implications for HIV prevention and treatment. AIDS Care. 2015;27(3):273-82.
- 55. Curioso WH, Quistberg DA, Cabello R, Gozzer E, Garcia PJ, Holmes KK, Kurth AE. "It's time for your life": How should we remind patients to take medicines using short text messages? AMIA Annu Symp Proc. 2009;2009:129-33.
- 56. Mugavero MJ, Westfall AO, Zinski A, Davila J, Drainoni ML, et al. Retention in Care (RIC) Study Group. Measuring retention in HIV care: the elusive gold standard. J Acquir Immune Defic Syndr. 2012 Dec 15;61(5):574-80.
- 57. Gardner EM, McLees MP, Steiner JF, Del Rio C, Burman WJ. The spectrum of engagement in HIV care and its relevance to test-and-treat strategies for prevention of HIV infection. Clin Infect Dis 2011; 52:793–800.
- 58. Yehia BR, Fleishman JA, Metlay JP, et al. Comparing different measures of retention in outpatient HIV care. AIDS 2012; 26:1131–9.

- 59. Van der Kop ML1, Karanja S, Thabane L, Marra C, Chung MH, Gelmon L, Kimani J, Lester RT. In-depth analysis of patient-clinician cell phone communication during the WelTel Kenya1 antiretroviral adherence trial. PLoS One. 2012;7(9):e46033.
- 60. Minick SG, May SB, Amico KR, Cully J, Davila JA, Kallen MA, Giordano TP. Participants' perspectives on improving retention in HIV care after hospitalization: A post-study qualitative investigation of the MAPPS study. PLoS One. 2018 Aug 27;13(8):e0202917.
- 61. Vagenas P, Brown SE, Clark JL, Konda KA, Lama JR, Sánchez J, Duerr AC, Altice FL. A Qualitative Assessment of Alcohol Consumption and Sexual Risk Behaviors Among Men Who Have Sex With Men and Transgender Women in Peru. Subst Use Misuse. 2017 Jun 7;52(7):831-839.
- 62. Braun V, Clarke V. Using thematic analysis in psychology. Qualitative Research in Psychology 2006; 3:77–101.
- 63. Creswell JW. (2012) Qualitative inquiry and research design: choosing among five approaches. New York: Sage Publications.
- 64. Mugavero MJ, Davila JA, Nevin CR, Giordano TP. From access to engagement: Measuring retention in outpatient HIV clinical care. AIDS Patient Care STDS 2010;24:607–613.
- 65. Technical Standard for Integral Attention of the Adult with Infection by the Human Immunodeficiency Virus (HIV). Peru, March 2018. Retrieved from: <a href="ftp://ftp2.minsa.gob.pe/normaslegales/2018/R.M">ftp://ftp2.minsa.gob.pe/normaslegales/2018/R.M</a> 215-2018-MINSA.PDF
- 66. Lester RT1. Ask, don't tell mobile phones to improve HIV care. N Engl J Med. 2013 Nov 7;369(19):1867-8.
- 67. Radloff, Lenore S. The CES-D Scale: A self-report depression scale for research in the general population. Applied Psychological Measurement. 1977; 1(3):385–401.
- 68. Judith B. Cornelius, Jacek Dmochowski, Cherrie Boyer, Janet St Lawrence, Marguerita Lightfoot, Michael Moore. Text-Messaging-Enhanced HIV Intervention for African American Adolescents: A Feasibility Study. J Assoc Nurses AIDS Care. 2013 May-Jun; 24(3): 256–267.
- 69. Saunders RP, Evans MH, Joshi P. Developing a process-evaluation plan for assessing health promotion program implementation: a how-to guide. Health Promot Pract. 2005 Apr;6(2):134-47.
- 70. Liu AY, Vittinghoff E, von Felten P, et al. Randomized Controlled Trial of a Mobile Health Intervention to Promote Retention and Adherence to Preexposure Prophylaxis Among Young People at Risk for Human Immunodeficiency Virus: The EPIC Study. Clin Infect Dis. 2019;68(12):2010–2017. doi:10.1093/cid/ciy810

- 71. Rodríguez-Morales AJ, Bonilla-Aldana DK, Morales M, Suárez JA, Martínez-Buitrago E. Migration crisis in Venezuela and its impact on HIV in other countries: the case of Colombia. Ann Clin Microbiol Antimicrob. 2019;18(1):9. Published 2019 Mar 8. doi:10.1186/s12941-019-0310-4
- 72. Rebolledo-Ponietsky K, Munayco CV, Mezones-Holguín E. Migration crisis in Venezuela: impact on HIV in Peru. J Travel Med. 2019 Feb 1;26(2). pii: tay155. doi: 10.1093/jtm/tay155.
- 73. Alcalde-Rabanal Jacqueline Elizabeth, Lazo-González Oswaldo, Nigenda Gustavo. Sistema de salud de Perú. Salud pública Méx [revista en la Internet]. 2011 Ene [citado 2019 Nov 05]; 53( Suppl 2 ): s243-s254. Disponible en: <a href="http://www.scielo.org.mx/scielo.php?script=sci\_arttext&pid=S0036-36342011000800019&lng=es">http://www.scielo.org.mx/scielo.php?script=sci\_arttext&pid=S0036-36342011000800019&lng=es</a>.
- 74. Kelsey et al., Methods in Observational Epidemiology 2nd Edition, Table 12-15 Fleiss, Statistical Methods for Rates and Proportions, formulas 3.18 &3.19.

# APPENDIX 1 INFORMED CONSENT FORM

# **Study Title:**

A mobile phone short message service intervention to increase retention in HIV care among HIV-positive men who have sex with men in Peru.

#### Investigators:

Luis Menacho, Giovani Díaz, Magaly Blas, Elsa Gonzáles

#### Institution:

Universidad Peruana Cayetano Heredia

#### Purpose of the study:

We are inviting you to participate in a study to see the usefulness of a new text message followup strategy to help you keep appointments at this care service, and to provide you with ongoing support. This is a study developed by researchers from the Universidad Peruana Cayetano Heredia and the Alexander Von Humboldt Institute of Tropical Medicine.

We have seen that as time goes by, many patients receiving antiretroviral treatment stop coming for some controls. As a consequence, their health status cannot be assessed, they do not collect their medications, and they run the risk that the therapy will no longer work as well. The objective of this study is to evaluate a new strategy to motivate them and remind them not to stop coming to their controls.

#### **Procedures:**

If you decide to participate in this study, the following will be done:

- 1. You will need to provide your cell phone number and email address.
- 2. You will need to complete an online survey at the beginning, middle (at 6 months) and at the end of the study (at 12 months). We will send this survey to you by mail or cell phone. It will last 30 minutes (32 short items) and you will be asked for brief demographic information, sexual behavior, attendance at check-ups, and about some of your physical and mental health habits.
- 3. Some participants will receive text messages from a health provider approximately once a week for 6 months. They will be informative messages, reminders and also motivating. For confidentiality, a neutral language will be used and some messages will be private: you will be able to see them only if you enter the password that you will be given at the beginning. You can reply to messages if you have any questions, or a member of the team will call you back if you need them.

#### Risks:

There is a possibility of a breach in confidentiality if someone else reads your cell phone. We will minimize this risk by sending text messages with neutral language that does not contain words directly related to HIV to anticipate if someone else reads the text messages on your cell phone. In addition, text messages with additional information will be protected by a password that only

you will know. We recommend having the cell phone with a password, which is very common now. There is a possibility that some of the questions in the follow-up online surveys may cause you some discomfort, you are free to answer them or not.

#### Benefits:

You may benefit from receiving informative, reminder and also motivational text messages to help you keep appointments, stay in care which will help maintain good health. Likewise, you could receive logistical and emotional support from health providers.

#### Costs and compensation

You will not have to pay anything to participate in the study. Likewise, you will not receive any economic or other incentive.

# Confidentiality:

We will store your information with codes and not with names. Only researchers will have access to the databases. If the results of this study are published, no information will be shown that allows the identification of the people who participated in this study.

# Participant rights:

If you decide to participate in the study, you may withdraw from the study at any time, or not participate in part of the study without harm. If you have any further questions, please ask the study staff or call Dr. Luis Menacho at 991671979.

If you have questions about the ethical aspects of the study, or believe that you have been treated unfairly, you can contact Dr. Frine Samalvides Cuba, president of the Institutional Research Ethics Committee of the Universidad Peruana Cayetano Heredia at telephone 01-3190000 annex 201355, the which will be enabled soon so, in the meantime, you can send an email to: <a href="mailto:duict.cieh@oficinas-upch.pe">duict.cieh@oficinas-upch.pe</a>

A copy of this informed consent will be provided to you.

#### **DECLARATION AND/OR CONSENT**

I voluntarily agree to participate in this study, I understand the activities I will participate in if I decide to enter the study, I also understand that I can decide not to participate and that I can withdraw from the study at any time.

| Name (participant):<br>Date and time: |
|---------------------------------------|
| Name (investigator) Date and time: |